CLINICAL TRIAL: NCT05243030
Title: Adapting Effective mHealth Interventions to Improve Uptake and Adherence of the HIV Pre-exposure Prophylaxis (PrEP) in Thai Young Men Who Have Sex With Men (MSM).
Brief Title: Developing mHealth to Promote PrEP Use Among Thai Young Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Wayne State University (Other); Institute of HIV Research and Innovation Foundation, Thailand (Other)
Responsible Party: Principal Investigator, Bo Wang, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H00023523; 1R34MH124081-01A1 (NIH)
Record Dates: First submitted 2022-01-18; First posted 2022-02-16 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Pre-Exposure Prophylaxis
Keywords: Pre-exposure Prophylaxis (PrEP); HIV Prevention; Mobile health (mHealth)

STUDY DESIGN:
Intervention Model Description: 2-arm RCT with 2:1 randomization to MES-PrEP+MTM or standard PrEP Counseling
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MES-PrEP and MTM (Experimental): Participants in this arm will receive standard PrEP counseling, followed by mHealth interventions to improve PrEP uptake and support PrEP adherence.
  Interventions: Behavioral: Motivational Enhancement System for PrEP Uptake and Adherence (MES-PrEP); Behavioral: Motivational Interactive Text Messaging (MTM); Behavioral: Standard PrEP Counseling
- Standard PrEP Counseling (Active Comparator): Participants in this arm will receive the standard PrEP counseling.
  Interventions: Behavioral: Standard PrEP Counseling

INTERVENTIONS:
Behavioral: Motivational Enhancement System for PrEP Uptake and Adherence (MES-PrEP) — MES-PrEP is a two-session computer-delivered intervention based on IMB model. The intervention is tailored based on the person's ratings of perceived importance and confidence of initiating PrEP and sustaining adherence to PrEP. Participants are routed to different intervention content based on their assessment of their importance and confidence. Youth are provided with feedback on scores on the knowledge assessment followed by information about protective effect that can result from improved PrEP adherence. Finally, participants are asked to set a goal: obtain PrEP prescription, optimal adherence, practice steps, or thinking about it more, and they form plans for overcoming barriers. In the second session, branches are based on whether the youth felt they met the goal, partially met the goal, or did not meet the goal. Sessions of MES-PrEP will occur at baseline and month 1.
  Arms: MES-PrEP and MTM
Behavioral: Motivational Interactive Text Messaging (MTM) — Participants will receive automated motivational text messages to promote PrEP initiation and adherence. These contents will be customized based on their readiness to change in regards to PrEP. The message content is individualized based on participant response to baseline survey. Those participants who indicate that they are "ready" to set the goal to take PrEP will receive text messages reminding them to take PrEP. Those who indicate that they are less than ready to take their PrEP can choose from a range of alternatives, such as taking on-demand PrEP or just think about taking PrEP. For those who are not ready to take PrEP, the content will be individualized based on the participant's choice, i.e., a daily message encouraging them to work toward their chosen goal. Participants who are currently not on PrEP will receive daily text messages regarding PrEP effectiveness, HIV risk and where to access PrEP.
  Arms: MES-PrEP and MTM
Behavioral: Standard PrEP Counseling — All participants will received one-on-one, face to face counseling from lay providers at baseline, months 1, 3 and 6. Standard PrEP counseling includes sexual and behavioral risk assessment for HIV/STIs and risk reduction. For those not on PrEP, the sessions will focus on risk perception, awareness of PrEP/post-exposure prophylaxis (PEP) and facilitators and barriers of accessing PrEP. For those on PrEP, the sessions will focus on adherence. Standard counseling sessions will be nonjudgmental, non-discriminatory and client-centered.

SUMMARY:
The goal of this study is to develop and pilot test technology-based interventions to promote Pre-exposure Prophylaxis (PrEP) uptake and adherence among Thai young men who have sex with men (YMSM).

DETAILED DESCRIPTION:
Motivational Enhancement System for Adherence (MESA) is a computer-based motivation invention, based on the Information-Motivation-Behavioral Skills (IMB) model and Motivational Interviewing (MI) principles, used to promote adherence among HIV-positive youth initiating antiretroviral treatment. In this study, the team will adapt and develop MESA to focus on PrEP uptake and adherence, which will be called Motivational Enhancement System for PrEP Uptake and Adherence (MES-PrEP). Motivational Interactive Text Messaging (MTM) will be integrated with MES-PrEP to provide ongoing support to maintain the individual's motivation for behavior change. Both interventions will be developed and refined based upon the inputs from YMSM through focus group discussion and youth advisory board.

The Investigators propose to pilot randomized controlled trial (RCT) to evaluate the feasibility, acceptability, and preliminary efficacy of an intervention combining MES-PrEP and MTM to increase PrEP uptake and adherence among Thai YMSM. Eligible YMSM will be randomized to receive either the intervention plus the standard PrEP counseling or standard PrEP counseling, and followed for 6 months with assessments at baseline, month 1, 3 and 6.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-25 years old
* Men who report sex with men in the past 12 months
* Confirmed HIV-negative status
* Self-reported evidence of being at-risk for HIV acquisition, including one of the following in the past 6 months:

  1. having a sex with an HIV-positive partner
  2. having anal sex
  3. without using a condom
  4. being diagnosed with an STI or
  5. having any illicit drug use (e.g., Amphetamine type stimulants)
* Able to understand, read and speak Thai
* Either having not started PrEP (Group 1: PrEP naive) or currently on PrEP but not adherent to PrEP (taking ≤3 pills/week) in the past month (Group 2: PrEP users).

Exclusion Criteria:

* In a mutually monogamous relationship of more than 6 months with a partner who recently tested HIV-negative
* Have a serious cognitive or psychiatric problem that would compromise ability to provide informed consent
* currently enrolled in another HIV intervention study

Ages: 16 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Men who have sex with men
Enrollment: 119 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Intervention Acceptability: System Usability Score | Month 3
  System Usability Score (SUS) is a 10-item, Likert scale used to calculate intervention usability. Each item ranges from 0 to 4 (with 4 being the most positive response). For odd-numbered items, the score is calculated by subtracting one from the user response. For even-numbered items, the score is calculated by subtracting the user response from 5. Then sum the total score and multiply that by 2.5. The overall SUS scores range from 0 to 100. A score of > 50 indicates that the technology-based interventions are acceptable.
Intervention Acceptability: System Usability Score | Month 6
  System Usability Score (SUS) is a 10-item, Likert scale used to calculate intervention usability. Each item ranges from 0 to 4 (with 4 being the most positive response). For odd-numbered items, the score is calculated by subtracting one from the user response. For even-numbered items, the score is calculated by subtracting the user response from 5. Then sum the total score and multiply that by 2.5. The overall SUS scores range from 0 to 100. A score of > 50 indicates that the technology-based interventions are acceptable.
Intervention Acceptability: Client Satisfaction Questionnaire | Month 3
  Client Satisfaction Questionnaire (CSQ-8) is an 8-items, Likert scale measuring the construct of global intervention satisfaction. The total possible composite score range from 8 to 32, with higher scores indicating a greater degree of acceptability.
Intervention Acceptability: Client Satisfaction Questionnaire | Month 6
  Client Satisfaction Questionnaire (CSQ-8) is an 8-items, Likert scale measuring the construct of global intervention satisfaction. The total possible composite score range from 8 to 32, with higher scores indicating a greater degree of acceptability.
Intervention Feasibility: Number of responses to text messages | Baseline through Month 6
  Intervention feasibility will be measured by total number of responses to text messages. Point estimates of >50% of participants responded to at least one text message is considered as the minimum criteria for feasibility.
Intervention Feasibility: Number of intervention sessions completed | Baseline through Month 6
  Intervention feasibility will be measured by number of intervention sessions completed. Point estimates of >50% of participants completed at least one intervention session is considered as the minimum criteria for feasibility.
Intervention Feasibility: Participant retention | Baseline through Month 6
  Intervention Feasibility will be measured by participants retention rate at Month 6.
PrEP Adherence: Visual analog scale | Baseline through Month 6
  PrEP adherence will be measured from Young Adult Adherence Interview via computer-assisted self-interview (CASI) survey which contains a visual analog scale (VAS). VAS ranges from 0 to 100, with higher percentage indicating greater adherence to PrEP.
PrEP Adherence: Self-reported adherence | Baseline through Month 6
  PrEP adherence will be measured from self-reported adherence to PrEP in the past 4 weeks.
PrEP Adherence: Dried blood spots | Baseline through Month 6
  PrEP adherence will be measured by the level of tenofovir in dried blood spots (DBS). DBS report on 80% Truvada adherence after at least three weeks of regular adherence.
PrEP uptake | Month 1 through Month 6
  PrEP uptake will be measured by the number of PrEP prescription, using a self-report measure (participants reporting if they left the clinic with PrEP) and confirming with clinic records.

SECONDARY OUTCOMES:
PrEP Knowledge | Baseline to Month 6
  Knowledge of PrEP will be measured using the 13-item PrEP knowledge scale. The total possible score is 13, with higher scores indicating a greater degree of PrEP knowledge.
HIV Knowledge | Baseline to Month 6
  Knowledge of HIV transmission risk will be assessed using am 18-item HIV Knowledge Questionnaire. The total possible composite score range from 0 to 18, with higher scores indicating a greater degree of HIV knowledge.
Motivation: Rollnick's Readiness Ruler | Baseline to Month 6
  Behavioral intentions will be measured using 5-item Rollnick's Readiness Ruler, which correspond to PrEP uptake and adherence. Each item ranges from 0 to 10, with higher numbers indicate greater readiness for change.
Motivation: Decisional Balance for PrEP Use | Baseline to Month 6
  Attitude towards PrEP will be measured using 36-item Decisional Balance for PrEP Use. The 5-point Likert scale assesses the pros and cons of PrEP use and is helpful in understanding cognitive and motivational aspects of decision making.
Behavioral Skill | Baseline to Month 6
  Behavior skills will be assessed using the 8-item adapted version of Self-Efficacy for Health Promotion and Risk Reduction Questionnaire. The 5-point Likert scale assesses the confidence in using a condom, taking PrEP as recommended and getting PrEP refills. The total possible score is 40, with higher scores indicating a greater confidence for each item.
HIV Status | Baseline to Month 6
  HIV status based on 4th generation HIV-1/2 antigen/antibody combo testing.
Sexually Transmitted Infections (STIs) Diagnosis | Baseline to Month 6
  STI diagnosis based on treponemal test with rapid plasma reagin (RPR) confirmation for syphilis. Pooled urine, oropharyngeal and rectal swabs for gonorrhea and chlamydia nucleic acid amplification test (NAAT) testing.
Sexual Risk | Baseline to Month 6
  Sexual risk will be assessed through Timeline Followback via CASI, which collects sexual behavior in the past 30 days, including questions about condom use and number of sexual partners.

OTHER OUTCOMES:
Mental Health | Baseline to Month 6
  Mental Health will be assessed using the 12-item Thai General Health Questionnaire. The 4-point Likert scale measures psychological distress such as depression, anxiety, social impartment and somatic complaints. All items are rated on a 4-point Likert scale. The total possible score is 48, with higher scores indicating higher severity of psychological distress.
PrEP-related Stigma | Baseline to Month 6
  PrEP-related stigma will be assessed using the 10-item PrEP stigma and positive attitudes scale. The 5-point Likert scale measures opinions about PrEP.
Social support | Baseline to Month 6
  Social support will be assessed using the 13-item Social Provision Scale (SPS). The 5-point Likert scale measures the availability of social support, including emotional support, information support, instrumental support, companionship and social isolation. The total possible score is 65, with higher scores indicating greater availability of social support.
Perceived HIV risk | Baseline to Month 6
  Perceived HIV risk will be measured using the 8-item Perceived Risk of HIV Scale. Higher scores indicating higher perceived risk for HIV.
Drug/Alcohol Use: ASSIST | Baseline to Month 6
  Drug/Alcohol Use will be assessed using Alcohol, Smoking and Substance Involvement Screening Test (ASSIST) developed by the World Health Organization (WHO). ASSIST is a questionnaire that is used for identification of substance use related health risks and substance use disorders. Each item ranges from 0-12, with 0 reflecting low risk score. The total possible score is 24, with higher number indicating higher risk of health and other problems based from the current pattern of substance use.
Drug/Alcohol Use: AUDIT-C | Baseline to Month 6
  Alcohol Use Disorders Identification Test (AUDIT-C) or a brief alcohol screening instrument will also be used to identify persons who are hazardous drinkers or have active alcohol use disorders (including alcohol abuse or dependence). Each item ranges from 0 to 4, with 0 reflecting no alcohol use. The total possible score is 12, with higher number indicating higher drink above recommended limits and are at increased risks for harm.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, PhD, Principal Investigator — University of Massachusetts, Worcester
Locations (3):
- Thailand (3):
  - Rainbow Sky Association of Thailand, Bangkok, Bangkok
  - Institute of HIV Research and Innovation, Bangkok, Bangkok
  - SWING Foundation, Bangkok, Bangkok

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected during the study, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Colby D, Srithanaviboonchai K, Vanichseni S, Ongwandee S, Phanuphak N, Martin M, Choopanya K, Chariyalertsak S, van Griensven F. HIV pre-exposure prophylaxis and health and community systems in the Global South: Thailand case study. J Int AIDS Soc. 2015 Jul 20;18(4 Suppl 3):19953. doi: 10.7448/IAS.18.4.19953. eCollection 2015. PMID 26198342
- [Background] Phanuphak N, Sungsing T, Jantarapakde J, Pengnonyang S, Trachunthong D, Mingkwanrungruang P, Sirisakyot W, Phiayura P, Seekaew P, Panpet P, Meekrua P, Praweprai N, Suwan F, Sangtong S, Brutrat P, Wongsri T, Na Nakorn PR, Mills S, Avery M, Vannakit R, Phanuphak P. Princess PrEP program: the first key population-led model to deliver pre-exposure prophylaxis to key populations by key populations in Thailand. Sex Health. 2018 Nov;15(6):542-555. doi: 10.1071/SH18065. PMID 30249317
- [Background] Naar-King S, Outlaw AY, Sarr M, Parsons JT, Belzer M, Macdonell K, Tanney M, Ondersma SJ; Adolescent Medicine Network for HIV/AIDS Interventions. Motivational Enhancement System for Adherence (MESA): pilot randomized trial of a brief computer-delivered prevention intervention for youth initiating antiretroviral treatment. J Pediatr Psychol. 2013 Jul;38(6):638-48. doi: 10.1093/jpepsy/jss132. Epub 2013 Jan 28. PMID 23359664
- [Background] Kolmodin MacDonell K, Naar S, Gibson-Scipio W, Lam P, Secord E. The Detroit Young Adult Asthma Project: Pilot of a Technology-Based Medication Adherence Intervention for African-American Emerging Adults. J Adolesc Health. 2016 Oct;59(4):465-71. doi: 10.1016/j.jadohealth.2016.05.016. Epub 2016 Jul 27. PMID 27475032
- [Background] Horvath T, Azman H, Kennedy GE, Rutherford GW. Mobile phone text messaging for promoting adherence to antiretroviral therapy in patients with HIV infection. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009756. doi: 10.1002/14651858.CD009756. PMID 22419345
- [Background] Thienkrua W, van Griensven F, Mock PA, Dunne EF, Raengsakulrach B, Wimonsate W, Howteerakul N, Ungsedhapand C, Chiwarakorn A, Holtz TH. Young Men Who Have Sex with Men at High Risk for HIV, Bangkok MSM Cohort Study, Thailand 2006-2014. AIDS Behav. 2018 Jul;22(7):2137-2146. doi: 10.1007/s10461-017-1963-7. PMID 29138981
- [Background] Wheelock A, Eisingerich AB, Ananworanich J, Gomez GB, Hallett TB, Dybul MR, Piot P. Are Thai MSM willing to take PrEP for HIV prevention? An analysis of attitudes, preferences and acceptance. PLoS One. 2013;8(1):e54288. doi: 10.1371/journal.pone.0054288. Epub 2013 Jan 14. PMID 23342121
- [Background] Seekaew P, Nguyen E, Sungsing T, Jantarapakde J, Pengnonyang S, Trachunthong D, Mingkwanrungruang P, Sirisakyot W, Phiayura P, Panpet P, Meekrua P, Praweprai N, Suwan F, Sangtong S, Brutrat P, Wongsri T, Nakorn PRN, Mills S, Avery M, Vannakit R, Phanuphak P, Phanuphak N. Correlates of nonadherence to key population-led HIV pre-exposure prophylaxis services among Thai men who have sex with men and transgender women. BMC Public Health. 2019 Mar 21;19(1):328. doi: 10.1186/s12889-019-6645-0. PMID 30898095
- [Background] Beyrer C, Baral SD, van Griensven F, Goodreau SM, Chariyalertsak S, Wirtz AL, Brookmeyer R. Global epidemiology of HIV infection in men who have sex with men. Lancet. 2012 Jul 28;380(9839):367-77. doi: 10.1016/S0140-6736(12)60821-6. Epub 2012 Jul 20. PMID 22819660
- [Background] Chan PA, Mena L, Patel R, Oldenburg CE, Beauchamps L, Perez-Brumer AG, Parker S, Mayer KH, Mimiaga MJ, Nunn A. Retention in care outcomes for HIV pre-exposure prophylaxis implementation programmes among men who have sex with men in three US cities. J Int AIDS Soc. 2016 Jun 13;19(1):20903. doi: 10.7448/IAS.19.1.20903. eCollection 2016. PMID 27302837
- [Background] Schnall R, Travers J, Rojas M, Carballo-Dieguez A. eHealth interventions for HIV prevention in high-risk men who have sex with men: a systematic review. J Med Internet Res. 2014 May 26;16(5):e134. doi: 10.2196/jmir.3393. PMID 24862459
- [Background] Parsons JT, Lelutiu-Weinberger C, Botsko M, Golub SA. A randomized controlled trial utilizing motivational interviewing to reduce HIV risk and drug use in young gay and bisexual men. J Consult Clin Psychol. 2014 Feb;82(1):9-18. doi: 10.1037/a0035311. Epub 2013 Dec 23. PMID 24364800
- [Background] Naar-King S, Outlaw A, Green-Jones M, Wright K, Parsons JT. Motivational interviewing by peer outreach workers: a pilot randomized clinical trial to retain adolescents and young adults in HIV care. AIDS Care. 2009 Jul;21(7):868-73. doi: 10.1080/09540120802612824. PMID 20024744
- [Background] Liu AY, Vittinghoff E, von Felten P, Rivet Amico K, Anderson PL, Lester R, Andrew E, Estes I, Serrano P, Brothers J, Buchbinder S, Hosek S, Fuchs JD. Randomized Controlled Trial of a Mobile Health Intervention to Promote Retention and Adherence to Preexposure Prophylaxis Among Young People at Risk for Human Immunodeficiency Virus: The EPIC Study. Clin Infect Dis. 2019 May 30;68(12):2010-2017. doi: 10.1093/cid/ciy810. PMID 30239620
- [Background] Dubov A, Altice FL, Fraenkel L. An Information-Motivation-Behavioral Skills Model of PrEP Uptake. AIDS Behav. 2018 Nov;22(11):3603-3616. doi: 10.1007/s10461-018-2095-4. PMID 29557540
- [Background] Badawy SM, Barrera L, Sinno MG, Kaviany S, O'Dwyer LC, Kuhns LM. Text Messaging and Mobile Phone Apps as Interventions to Improve Adherence in Adolescents With Chronic Health Conditions: A Systematic Review. JMIR Mhealth Uhealth. 2017 May 15;5(5):e66. doi: 10.2196/mhealth.7798. PMID 28506955
- [Background] Rongkavilit C, Naar-King S, Kaljee LM, Panthong A, Koken JA, Bunupuradah T, Parsons JT. Applying the information-motivation-behavioral skills model in medication adherence among Thai youth living with HIV: a qualitative study. AIDS Patient Care STDS. 2010 Dec;24(12):787-94. doi: 10.1089/apc.2010.0069. Epub 2010 Nov 22. PMID 21091238
- [Background] van Griensven F, Varangrat A, Wimonsate W, Tanpradech S, Kladsawad K, Chemnasiri T, Suksripanich O, Phanuphak P, Mock P, Kanggarnrua K, McNicholl J, Plipat T. Trends in HIV Prevalence, Estimated HIV Incidence, and Risk Behavior Among Men Who Have Sex With Men in Bangkok, Thailand, 2003-2007. J Acquir Immune Defic Syndr. 2010 Feb;53(2):234-9. doi: 10.1097/QAI.0b013e3181c2fc86. PMID 19901844
- [Background] Dowshen N, Kuhns LM, Johnson A, Holoyda BJ, Garofalo R. Improving adherence to antiretroviral therapy for youth living with HIV/AIDS: a pilot study using personalized, interactive, daily text message reminders. J Med Internet Res. 2012 Apr 5;14(2):e51. doi: 10.2196/jmir.2015. PMID 22481246
- [Background] Yu YJ, Schieber E, Janamnuaysook R, Wang B, Gunasekar A, MacDonell K, Getwongsa P, Kim D, Wongharn P, Phanuphak N. Barriers and facilitators to pre-exposure prophylaxis (PrEP) uptake and adherence among men who have sex with men (MSM) in Thailand: a qualitative study. AIDS Care. 2024 Aug;36(8):1126-1134. doi: 10.1080/09540121.2024.2332443. Epub 2024 Apr 4. PMID 38574278
- [Derived] Wang B, Janamnuaysook R, MacDonell K, Rongkavilit C, Schieber E, Naar S, Phanuphak N. Adapting Effective mHealth Interventions to Improve Uptake and Adherence to HIV Pre-Exposure Prophylaxis Among Thai Young Men Who Have Sex With Men: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Sep 4;12:e46435. doi: 10.2196/46435. PMID 37665622